CLINICAL TRIAL: NCT01882452
Title: A Randomised Controlled Clinical Trial of Memory Specificity Training (MEST) for Depression
Acronym: MEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Professor Tim Dalgleish, Professor, Medical Research Council
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEST-UK
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder; Depressive Symptoms
Keywords: Memory specificity training; Autobiographical memory; Major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Educational Status; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memory Specificity Training (Experimental): Five weekly one-hour sessions of memory specificity training administered in groups of 5-8 participants.
  Interventions: Behavioral: Memory Specificity Training
- Education and Support (Active Comparator): Five weekly one-hour sessions of an education-and-discussion supportive intervention, administered in groups of 5-8 participants.
  Interventions: Behavioral: Education and Support

INTERVENTIONS:
Behavioral: Memory Specificity Training — This intervention is a manualised, structured treatment delivered over 5 x 60 minute sessions to groups of 5-8 individuals. This treatment involves repeated practice of retrieving specific autobiographical memories in response to positive, negative and neutral cue words. There is a single psychoeducation component in the first session about memory difficulties common in depression which provides the rationale for this treatment. The training is supplemented by weekly homework practice.
  Arms: Memory Specificity Training
Behavioral: Education and Support — The education-and-support comparison condition is matched with the experimental arm for length and format (ie., 5 x 60 minute weekly sessions in groups of 5-8 individuals). Groups receive a single psychoeducation component where information about depression is provided. This is followed by non-directive support where participants are encouraged to raise different kinds of events that occur each week for discussion in the group. The sessions are supplemented by a homework diary where participants will be invited to note down an event that occurs each day, which may be positive, negative, or benign and non-emotional in nature. This material will provide the basis for discussion in the weekly group meetings.
  Arms: Education and Support

SUMMARY:
Depression involves the tendency to recall overgeneral personal memories, a phenomenon which has been linked to numerous adverse psychological outcomes. The purpose of this study is to investigate whether a group-based Memory Specificity Training (MEST) programme improves outcomes in depression, and how this compares to an education and support control group. The primary aim is to examine whether MEST, which involves repeated practice retrieving specific autobiographical memories reduces depressive symptoms immediately post-treatment, and whether this is maintained 3 months after treatment. The secondary objective of this trial is to examine the role of hypothesised cognitive processes (ie., rumination, executive control, cognitive avoidance) which may underlie improvements in depression and memory.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of Major Depressive Disorder
* History of more than one previous depressive episode
* Current diagnosis of a Major Depressive Episode
* Depressive symptoms rated in the mild-severe range (> 13 on the BDI-II)
* Memory specificity < .70 (as assessed on the AMT)

Exclusion Criteria:

* Head trauma
* Organic brain damage
* Secondary diagnosis of another affective disorder
* Psychosis
* Current drug or alcohol abuse or dependence
* A diagnosed Axis II disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms on the Beck Depression Inventory II (BDI-II) | Change from baseline to 3 months post-treatment
  Symptom severity score

SECONDARY OUTCOMES:
Change in depressive status according to the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders - IV (SCID-IV) | Change from baseline at end of treatment (approximately 6 weeks) and 3 months post-treatment, and 6-months post-treatment (6-month follow-up for MEST group only)
  Presence of a current Major Depressive Episode (MDE)
Change from baseline in autobiographical memory specificity on Autobiographical Memory Test (AMT) | Change from baseline at end of treatment (approximately 6 weeks) and 3 months post-treatment
  Memory specificity level
Change from baseline in depressive symptoms as measured on the BDI-II | Change from baseline to post-treatment (approximately 6-weeks)
  Symptom severity score
Depression free days following treatment according to the Longitudinal Follow-up Evaluation on the SCID-IV | Post-treatment and 3-month and 6-month follow-up
  Number of depression-free days

OTHER OUTCOMES:
Change from baseline on the Beck Anxiety Inventory (BAI) | Change from baseline at end of treatment (approximately 6 weeks) and 3 months post-treatment
  Symptom severity score
Change from baseline on the Beck Hopelessness Scale (BHS) | Change from baseline at end of treatment (approximately 6 weeks) and 3 months post-treatment
  Hopelessness score
Change from baseline on the Cognitive Avoidance Questionnaire (CAQ) | Change from baseline at end of treatment (approximately 6 weeks) and 3 months post-treatment
  Tendency for avoidance score
Change in baseline on Rumination Response Scale (RRS) | Change from baseline at end of treatment (approximately 6 weeks) and 3 months post-treatment
  Tendency to ruminate score
Change from baseline in performance on Means-Ends Problem Solving Task (MEPS) | Change from baseline at end of treatment (approximately 6 weeks) and 3 months post-treatment
  Problem solving effectiveness score
Change from baseline in performance on Verbal Fluency Task | Change from baseline at end of treatment (approximately 6 weeks) and 3 months post-treatment
  Index of executive control
Change in baseline on performance on Digit Span Task | Change from baseline at end of treatment (approximately 6 weeks) and 3 months post-treatment
  Working memory index

CONTACTS AND LOCATIONS:
Overall Officials: Tim Dalgleish, PhD, Principal Investigator — Medical Research Council
Locations (1):
- Aliza Werner-Seidler, Sydney, Australia

REFERENCES:
- [Derived] Werner-Seidler A, Hitchcock C, Bevan A, McKinnon A, Gillard J, Dahm T, Chadwick I, Panesar I, Breakwell L, Mueller V, Rodrigues E, Rees C, Gormley S, Schweizer S, Watson P, Raes F, Jobson L, Dalgleish T. A cluster randomized controlled platform trial comparing group MEmory specificity training (MEST) to group psychoeducation and supportive counselling (PSC) in the treatment of recurrent depression. Behav Res Ther. 2018 Jun;105:1-9. doi: 10.1016/j.brat.2018.03.004. Epub 2018 Mar 15. PMID 29587159
- [Derived] Dalgleish T, Bevan A, McKinnon A, Breakwell L, Mueller V, Chadwick I, Schweizer S, Hitchcock C, Watson P, Raes F, Jobson L, Werner-Seidler A. A comparison of MEmory Specificity Training (MEST) to education and support (ES) in the treatment of recurrent depression: study protocol for a cluster randomised controlled trial. Trials. 2014 Jul 22;15:293. doi: 10.1186/1745-6215-15-293. PMID 25052061